CLINICAL TRIAL: NCT03245177
Title: A Phase I Study of Pembrolizumab Anti PD-1 Monoclonal Antibody in Combination With Radiotherapy in Locally Advanced Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Pembrolizumab in Combination With Radiotherapy in Locally Advanced Non-Small Cell Lung Cancer (NSCLC)
Acronym: PARIS
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Funding withdrawn.
Sponsor: Prof Corinne Faivre-Finn (Other)
Collaborators: University of Leeds (Other); Merck Sharp & Dohme LLC (Industry); Cancer Research UK (Other)
Responsible Party: Sponsor-Investigator, Prof Corinne Faivre-Finn, Professor of Thoracic Radiation Oncology & Honorary Consultant Clinical Oncology, The Christie NHS Foundation Trust
Organization: The Christie NHS Foundation Trust (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CFTSp103
Record Dates: First submitted 2017-07-13; First posted 2017-08-10 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab plus radiotherapy (Experimental): Pembrolizumab is given by intravenous infusion over 30 minutes at a maximum dose of 200mg. The first dose of pembrolizumab is administered 14 days prior to the initiation of radiotherapy and every 3 weeks thereafter. Radiotherapy is given as a standard dose (60-66 Gy in 2 Gy/fraction) over 40-45 days (daily on Mon-Fri) Following completion of radiotherapy, participants will continue to receive pembrolizumab every 3 weeks for up to 12 months of maintenance treatment.
  Interventions: Biological: Pembrolizumab; Radiation: Radiotherapy

INTERVENTIONS:
Biological: Pembrolizumab — Anti-PD-1 antibody
Radiation: Radiotherapy — 60-66 Gy in 30-33 fractions, 2 Gy per fraction

SUMMARY:
Lung cancer is the leading cause of cancer mortality worldwide and in the U.K alone; there are 38,000 new cases of non-small cell lung cancer (NSCLC) a year. The new treatment being tested in this study is called pembrolizumab, this is a type of immunotherapy, which works by stimulating the body's own immune system to fight cancer cells.

Pembrolizumab blocks a protein on the T-cell surface (one of the cells of the immune system), which then triggers the cell to find and kill cancer cells. This will be given with radiotherapy to see if this combination is safe and effective at treating patients with non-small cell lung cancer.

Pembrolizumab has proved to be a safe and effective treatment for other cancers such as melanoma and lung cancer. Radiotherapy is often given as standard treatment to treat lung cancer, and is proven to be a safe and tolerable treatment. However, the safety of the combination of Pembrolizumab and thoracic radiotherapy delivered concurrently has not been tested yet prospectively

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed NSCLC
* Unresectable stage III NSCLC not suitable for concurrent chemoradiotherapy i.e;

  * Patient unsuitable for cisplatin (eg poor renal function);
  * Large volume of disease with predicted dose to thoracic organs at risk that are likely to exceed the constraints for concurrent chemoradiotherapy, in the opinion of a clinical oncologist specialised in lung cancer
* Stage IV NSCLC with dominant chest symptoms and low burden of metastatic disease who may benefit from thoracic RT
* Patient considered suitable for radical radiotherapy
* If chemotherapy has been given previously, the maximum interval between the last day of chemotherapy and the start of radiotherapy must be 6 weeks. The minimum interval between the last day of chemotherapy and the start of Pembrolizumab must be one week
* Age ≥ 18
* Life expectancy estimated to be greater than 6 months
* Performance status (ECOG) 0 or 1 (see Appendix 1)
* MRC dyspnoea score < 3 (see Appendix 2)
* FEV1 ≥ 40% predicted and DLCO ≥ 40% predicted; Lung V20 ≤ 30% in the dose finding part of the study and ≤ 35% in the expanded cohort
* No prior thoracic radiotherapy (excluding patients that have had RT for Breast cancer providing that the overlap is minimal as per local investigators discretion or as discussed and agreed by CI as required) or T cell modulating antibodies (including anti-PD-1, anti-PD-L1, PD-L2, anti-CD137 and anti-CTLA4, including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways)
* Measurable disease based on RECIST 1.1
* Patient willing to undergo a repeat biopsy post RT
* Written informed consent must be given according to GCP and national regulations.
* Adequate organ function within 7 days of study treatment as defined in the protocol.

Exclusion Criteria:

* Mixed non-small cell and small cell tumours
* Participation in a study of an investigational agent or using an investigational device within 4 weeks prior to the anticipated start of treatment.
* Current or previous malignant disease within 3 years except CIN, non-melanoma skin cancer and low grade, low stage prostate cancer found as incidental finding and not requiring treatment
* History of interstitial pneumonitis (to include diffuse alveolar damage, non-malignant causes of pneumonitis, acute respiratory distress syndrome, alveolitis, cryptogenic organising pneumonia, obliterative bronchiolitis, non-malignant causes of pulmonary fibrosis)
* Presence of brain metastases confirmed by CT or MR brain (unless suitable for local treatment such as SRS or Neurosurgery)
* History of autoimmune disease requiring steroids or immunosuppressive medication
* Uncontrolled hypothyroidism or hyperthyroidism
* Other diseases requiring immunosuppressive therapy greater than 28 days prior to the anticipated first dose of trial treatment.
* Other diseases requiring systemic glucocorticoid (doses <=10 mg prednisolone or equivalent) prior to the first dose of trial treatment.
* Received a prior autologous or allogeneic organ or tissue transplantation.
* Chronic GI disease likely to interfere with protocol treatment.
* Testing positive for human immunodeficiency virus, active hepatitis B or C infection.
* Treatment with live vaccine within 30 days prior to the first dose of trial treatment.
* Patients of reproductive potential who are unable to comply with effective contraception if sexually active during the study and for up to 120 days after the last dose of Pembrolizumab
* Women who are pregnant or breastfeeding. Women of childbearing potential must have a negative serum or urine pregnancy test
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-08 (Estimated); Primary Completion 2019-08-01 (Estimated); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Recommended phase II dose (RP2D) | Within the period from the start of treatment until 12 weeks after completion of combined pembrolizumab and thoracic radiotherapy
  The dose level at which < 2/6 participants experience dose limiting toxicity (DLT).
Dose limiting toxicity | Within the period from the start of treatment until 12 weeks after completion of combined pembrolizumab and thoracic radiotherapy.
  Non-haematologic:
  Any ≥grade 3 non-haematological toxicity definitely, probably or possibly related to the combination of Pembrolizumab and thoracic radiotherapy including:
  * Increased MRC dyspnoea score >2 grades from baseline or CTCAE dyspnoea grade ≥3 persisting for >7 days
  * Pneumonitis grade ≥4, or grade ≥3 persisting for >7 days despite optimal medical management.
  * Oesophagitis grade ≥4, or ≥3 persisting for >7 days despite optimal medical management
  * Toxicity leading to interruption of radiotherapy for >4 days. Any grade 4 toxicity that has not previously been reported with pembrolizumab and is considered at least possibly related to the combination of pembrolizumab with radiotherapy
  Haematologic:
  * Neutropenia ≥grade 3 with fever >38.5
  * Thrombocytopaenia ≥grade 4.
  Any other event, in the opinion of the Safety Review Committee, is considered to be clinically significant and related to trial treatment.

SECONDARY OUTCOMES:
Safety profile, based on the occurrence of SAEs, SARs and SUSARs | Until 90 days after participant completes study treatment. Assessed up to 17 months.
Toxicity profile, based on the occurrence of adverse events, as assessed by CTCAE v4.0 | Until 30 days after participant completes study treatment. Assessed up to 15 months.
Treatment compliance of Pembrolizumab combined with thoracic RT | Until end of treatment for each participant.
Best overall response to Pembrolizumab combined with thoracic RT (RECIST) | Assessed for each participant from the start of the treatment until disease progression/recurrence. Assessed up to 15 months
Best overall response to Pembrolizumab combined with thoracic RT (immune-related response | Assessed for each participant from the start of the treatment until disease progression/recurrence. Assessed up to 15 months
Progression Free survival | Calculated for each participant from the date of registration to first documented evidence of disease progression or death. Assessed up to 15 months.
  Participants who have not progressed at the time of analysis will be censored at the last date they were known to be alive and progression free.
Overall survival | Calculated for each participant from the date of registration to death. Assessed up to 15 months.
  Participants who have not died at the time of analysis will be censored at the last date they were known to be alive.

OTHER OUTCOMES:
Baseline biopsy expression level of the immunological checkpoint PD-L1 | Assessed for each participant at time of registration to the trial
Change in PD-L1 expression level following Pembrolizumab combined with thoracic RT | Assessed for each participant from the start of the treatment until disease progression/recurrence. Assessed up to 15 months
Immune monitoring of primary tumour and peripheral blood mononuclear cells | Assessed for each participant from the start of the treatment until disease progression/recurrence. Assessed up to 15 months

CONTACTS AND LOCATIONS:
Overall Officials: Corinne Faivre-Finn, Principal Investigator — The Christie NHS Foundation Trust and the University of Manchester

IPD SHARING:
Plan to Share IPD: No